CLINICAL TRIAL: NCT00218491
Title: A Controlled Trial of N-Acetylcysteine (NAC) for Cocaine Dependence
Brief Title: Effectiveness of N-Acetylcysteine (NAC) in Treating Cocaine Dependent Individuals - 1
Acronym: NAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Malcolm, Professor of Psychiatry, Family Medicine & Pediatrics, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-19903-1; R01DA019903 (NIH); R01-19903-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1200mg N-Acetylcysteine (Experimental): 1200mg N-Acetylcysteine
  Interventions: Drug: N-Acetylcysteine
- 2400mg N-Acetylcysteine (Experimental): 2400mg N-Acetylcysteine
  Interventions: Drug: N-Acetylcysteine
- Matching Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — 1200mg N-Acetylcysteine
  Arms: 1200mg N-Acetylcysteine
Drug: N-Acetylcysteine — 2400mg N-Acetylcysteine
  Arms: 2400mg N-Acetylcysteine
Drug: Matching Placebo — Matching Placebo
  Arms: Matching Placebo

SUMMARY:
Currently, no effective drug treatment exists for cocaine dependence. Glutamate levels are disrupted with long-term cocaine use. N-acetyl cysteine (NAC) is a drug that is metabolized by the body to form cysteine, an active compound that normalizes glutamate levels. The purpose of this study is to determine the safety and effectiveness of NAC in treating cocaine dependent individuals.

DETAILED DESCRIPTION:
Currently, no effective pharmacological treatment exists for cocaine dependence. Long-term use of cocaine disrupts normal glutamate levels. If addicts stop using cocaine, glutamate levels drop, which encourages addicts to continue seeking the drug. NAC is a drug that increases intracellular cysteine levels, which in turn leads to normalization of glutamate levels. Currently, NAC is used for the treatment of cystic fibrosis, heart disease, and acetaminophen overdose. Since NAC has the capability of restoring normal glutamate levels, it holds potential as a treatment for cocaine dependence. The purpose of this study is to determine the safety and effectiveness of NAC in treating cocaine dependent individuals. In addition, this study will evaluate cocaine craving and withdrawal symptoms in individuals taking NAC.

Participants in this double-blind, placebo-controlled trial will be randomly assigned to receive either NAC or placebo. All participants will undergo an initial evaluation, which will include a physical examination, an electrocardiogram, blood samples, urine tests, and cue reactivity measures. Participants in the NAC group will receive either 600 mg or 1200 mg of NAC, two times each day for 8 weeks. In addition, all participants will receive cognitive behavioral therapy throughout the study on a weekly basis. Cocaine use will be confirmed by a urine drug screen test, three times each week. Participants will be assessed on a number of biomedical and psychosocial variables known to influence cocaine treatment outcomes. After Week 2, participants will repeat the cue reactivity procedures, which will include measuring a participant's craving response when exposed to conditioned reminders of prior cocaine use.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cocaine dependence, as determined by a mini-SCID interview
* Currently dependent on cocaine
* Seeking treatment for cocaine abuse at the time of study entry
* Currently uses cocaine by smoking, nasal, or intravenous route of administration.
* Stable physical and mental health, as judged by an interview and physical examination
* If female, demonstrates a negative pregnancy test and agrees to use an adequate method of contraception for the duration of the study
* Lives within a 50 mile radius of the research program center and has reliable transportation

Exclusion Criteria:

* Meets DSM-IV criteria for dependence on any psychoactive substance other than cocaine, alcohol, nicotine, or marijuana
* Physiological dependence on alcohol, which requires medical detoxification
* History of significant liver, kidney, endocrine, cardiac (e.g., arrhythmia requiring medication, angina pectoris, myocardial infarction), stroke, seizure, neurological, non-drug-related psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders (e.g., homocystinuria)
* History of an adverse reaction to cocaine, including loss of consciousness, chest pain, psychosis, or seizure
* History of adverse reaction or hypersensitivity to N-acetyl cystine (NAC), or a similar drug
* Significant active medical or psychiatric illness that might inhibit the ability to complete the study
* Active high blood pressure, defined as a mean of three sitting blood pressure readings of 145/95 or higher within a 10-day period
* History of or current asthma
* Occasional or daily use of albuterol or other beta-agonist inhalers
* Use of carbamazepine, phenytoin, nitrous oxide, methotrexate, 6 azauridine triacetate, or nitroglycerin within the 2 weeks prior to study entry
* Use of very large doses of folate, cyanocobalamine (vitamin B12), or pyridoxine (vitamin B6) as prescribed by a health care professional; individuals taking very large doses of these vitamins on a self-initiated basis may enter the study if they are willing to stop use 14 days prior to study entry and to use a standard generic multiple vitamin instead
* Pregnant or breastfeeding
* Required by the court to obtain treatment for cocaine dependence
* Not seeking treatment for cocaine dependence
* Anticipating elective surgery or hospitalization within 20 weeks of study entry
* Failure to have a consistent residence for the 4 weeks prior to study entry
* History of childhood or adult seizures
* Participated in cocaine treatment (clinical or research) within 30 days of study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malcolm, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1200mg N-Acetylcysteine | 2400mg N-Acetylcysteine | Matching Placebo
Started | 40 | 33 | 38
Completed | 40 | 33 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1200mg N-Acetylcysteine | 2400mg N-Acetylcysteine | Matching Placebo | Total
Number analyzed (Participants) | 40 | 33 | 38 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.1) | 43.3 (13.6) | 42.8 (8.7) | 43.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 10 | 28
  Male | 30 | 25 | 28 | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved Study Compliance
Description: Drug and placebo compliance were measured by urine riboflavin levels. Study compliance was defined as 80% or greater weekly urine riboflavin levels equal to or greater than 1500 ng/ml
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1200mg N-Acetylcysteine | 2400mg N-Acetylcysteine | Matching Placebo
Number analyzed (Participants) | 40 | 33 | 38
Participants | 22 | 15 | 18

ADVERSE EVENTS:
Arm/Group | 1200mg N-Acetylcysteine | 2400mg N-Acetylcysteine | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/33 | 0/38
Other Adverse Events (participants affected / at risk) | 32/40 | 28/33 | 28/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1200mg N-Acetylcysteine (N=40) | 2400mg N-Acetylcysteine (N=33) | Matching Placebo (N=38)
Change in Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatological episode (Skin and subcutaneous tissue disorders) | 5 (8) | 4 (4) | 2 (2)
Fall (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fever (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
GI Event (Gastrointestinal disorders) | 19 (29) | 20 (28) | 16 (23)
Respiratory event (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 7 (8)
Sleepiness (General disorders) | 1 (1) | 4 (5) | 2 (2)
Urinary disorder (Renal and urinary disorders) | 2 (3) | 2 (3) | 2 (2)
Muscle and Joint Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 5 (5)
Hyperactivity (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2)
Headache (General disorders) | 3 (4) | 3 (3) | 9 (11)
Insomnia (General disorders) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes